CLINICAL TRIAL: NCT04921800
Title: Feasibility Assessment of A Novel Wearable Skin Sensor for Post-Operative Monitoring Following Anterior Cervical Discectomy and Fusion (ACDF)
Brief Title: Measuring Dysphagia After ACDF Surgery Through A Novel Wearable Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STU00213413
Record Dates: First submitted 2021-03-05; First posted 2021-06-10 (Actual); Results first posted 2024-04-10 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2024-03

CONDITIONS: Cervical Spine Fusion
Keywords: cervical spine; fusion; discectomy; wearable technology
MeSH Terms: conditions — Klippel-Feil Syndrome | interventions — Gene Fusion

STUDY DESIGN:
Intervention Model Description: Patients enrolled in the study & scheduled for surgical intervention with anterior cervical discectomy and fusion will have the superficial sensor applied to the suprasternal notch following closure of the surgical incision. The data collected by the sensor will be recorded via a remote application and the sensor will then be removed 24 hours following placement. All patients enrolled in the study will be affixed with an identical sensor in accordance with the procedure outlined in the study protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Wearable Sensor Applied (Experimental): For these participants, the wearable ADAM sensor will be placed in the sternal notch to record anatomical data during the post-surgical period for up to 14 days
  Interventions: Procedure: Anterior Cervical Discectomy & Fusion; Device: Application of ADAM mechanoacoustic skin sensor

INTERVENTIONS:
Procedure: Anterior Cervical Discectomy & Fusion — Participants are undergoing previously scheduled anterior cervical discectomy & fusion for single level or multiple level cervical disease
Device: Application of ADAM mechanoacoustic skin sensor — Applying the ADAM sensor to the suprasternal notch following surgery to allow for collection of the anatomical data

SUMMARY:
The purpose of this study is to assess the function and reliability of a noninvasive, skin-like electronic sensor. The investigators hypothesize that this skin sensor will address an unmet need to wirelessly and noninvasively monitor and characterize the recovery process in post-operative patients who have undergone anterior cervical discectomy and fusion (ACDF). Specifically, the investigators will validate the use of the sensor in this patient population through monitoring of key physiological signals in the recovery process, including heart rate, respiratory rate, swallow count, talking time, energy expenditure, neck specific motion, and body orientation.

DETAILED DESCRIPTION:
Dysphagia, dysphonia, and loss of cervical range of motion (ROM) are common complications after anterior cervical spine surgery, specifically anterior cervical discectomy and fusion (ACDF). Despite their clinical importance, studies on the treatment and/or prevention of these complications are limited due to the lack of valid and reliable outcome measures. The majority of research is found in the otolaryngology literature and has focused on disease pathophysiology, diagnosis, and therapy.

Dysphagia and dysphonia are widely measured by patient self-reported questionnaires, including the MD Anderson Dysphasia Inventory and SWAL-QOL. However, these validated outcome tools are cumbersome to complete and, therefore, have not been widely accepted into clinical practice, including in postoperative ACDF patients. The Bazaz score, a subjective questionnaire that has not been validated in the literature, has also been used to evaluate dysphagia after ACDF. Assessment using the Bazaz score is based on clinical examination, with the surgeon listening to the patient's voice and documenting hoarseness in the post-operative period. Recently, new patient-centered outcomes, the Eating Assessment Tool (EAT-10) and Voice Handicap Index (VHI-10) have been developed. Both EAT-10 and VHI-10 have excellent validity and reliability in evaluating dysphagia and dysphonia, respectively, in post-operative ACDF patients and can be used to document the initial dysphagia or dysphonia severity and monitor the treatment response in people with a wide array of swallowing and voice disorders. However, these methods of evaluating dysphagia and dysphonia alone offer limited information about the severity and characteristic of dysphagia or dysphonia and do not provide continuous monitoring of swallowing or speaking function throughout the post-operative period.

The wearable sensors under investigation in this study offer a novel, noninvasive, and easy-to-use way to monitor dysphagia, dysphonia, cervical ROM, and overall recovery progress in post-operative ACDF patients. Previous testing has demonstrated the ability of our sensors to monitor vital signs (including heart rate and respiratory rate), swallow count, talking time, energy expenditure, cervical neck movement, and body orientation. Sensor-measured swallow count and talking time, in conjunction with EAT-10 and VHI-10 scores, can provide a comprehensive view of the progression of dysphagia and dysphonia. Cervical neck movements measured by the sensor can enable continuous assessment of cervical ROM. Other general metrics captured by the sensors, including heart rate, respiratory rate, energy expenditure, and body orientation can provide other meaningful measures of recovery in post-operative ACDF patients. These sensors have also received positive feedback from patients and physicians on their comfort, ease of use, and application, further demonstrating the potential value of these sensors in improving the quality of post-operative care for ACDF patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone anterior cervical discectomy and fusion (ACDF) for one or more levels for a diagnosis of cervical radiculopathy or myelopathy
* Scheduled to return to the MSK orthopaedic clinic for a post-operative appointment
* Aged between 18 to 88 years at time of surgery

Exclusion Criteria:

* Patients that underwent a revision of previous ACDF surgery at one or more operative levels
* Surgeries performed for a traumatic or oncologic etiology
* Members of vulnerable populations (i.e. prisoners, pregnant women)

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2024-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shuai Xu, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Wearable Sensor Applied
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Wearable Sensor Applied
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Vibrational Frequency of Vocalization Following Surgery
Description: Sensitivity of the device to mechanoacoustic output from motion and vocalization in hertz (Hz)
Time Frame: 0 to 24 hours post operative
Population: Investigators did not collect this variable.
Arm/Group | Wearable Sensor Applied
Number analyzed (Participants) | 0

2. Primary Outcome: Skin Temperature of the Surgical Site
Description: Sensitivity of the device to temperature of the surgical site in degrees Celsius
Time Frame: 0 to 24 hours post operative
Population: Investigators did not collect this variable.
Arm/Group | Wearable Sensor Applied
Number analyzed (Participants) | 0

3. Primary Outcome: Muscular Force Generated During Range of Motion Exercises
Description: Force vectors measured in gravitational acceleration units (g; 9.81 meters per second squared)
Time Frame: 0 to 24 hours post operative
Population: Investigators did not collect this variable.
Arm/Group | Wearable Sensor Applied
Number analyzed (Participants) | 0

4. Primary Outcome: Algorithm Validation
Description: Measuring the accuracy of the algorithm created to measure neck motion using the ADvanced Acousto-Mechanic sensor. Data analysis made no distinction between motion samples collected immediately after awaking from sedation in the post-anesthesia care unit and those collected immediately prior to discharge
Time Frame: Immediately after awaking from sedation in the post-anesthesia care unit and immediately prior to discharge
Population: patients
Measure: Mean (Standard Deviation); unit: percentage of correct motions detected
Arm/Group | Wearable Sensor Applied
Number analyzed (Participants) | 5
percentage of correct motions detected | 67.5 (5.8)

ADVERSE EVENTS:
Time Frame: 2 weeks postoperative
Arm/Group | Wearable Sensor Applied
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 5/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wearable Sensor Applied (N=11)
Pain (Musculoskeletal and connective tissue disorders) | 5 (5) — Patient was in too much pain to wear sensor and/or perform range of motion activities

LIMITATIONS AND CAVEATS:
The data collected by investigators did not match the a priori variables defined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT04921800/Prot_000.pdf
  • Informed Consent Form (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/00/NCT04921800/ICF_001.pdf